CLINICAL TRIAL: NCT03099616
Title: Automated Closed Loop Propofol Anaesthesia Versus Desflurane Inhalation Anaesthesia In Obese Patients Undergoing Bariatric Surgery: A Comparative Randomized Analysis of Recovery Profile
Brief Title: Automated Closed Loop Propofol Anaesthesia Versus Desflurane Inhalation Anaesthesia In Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Nitin Sethi (Other)
Responsible Party: Sponsor-Investigator, Dr Nitin Sethi, Doctor & Associate Professor, Sir Ganga Ram Hospital
Organization: Sir Ganga Ram Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EC/01/17/1105
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia; Bariatric Surgery
Keywords: propofol; CLADS; Desflurane; Obesity
MeSH Terms: conditions — Obesity | interventions — Propofol; Desflurane

STUDY DESIGN:
Intervention Model Description: 40 patients belonging to ASA physical patients status II and III of either sex, scheduled to undergo laparoscopic/robotic bariatric surgery (sleeve gastrectomy, Rouxen- Y gastric bypass) under general anaesthesia. The patients will be randomly allocated by computer generated numbers to one of the following two groups of 20 patients each.
  Group-1 [CLADS Group, n=20]: Anaesthesia will be induced and maintained with Propofol administered using the automated CLADS.
  Group-2 [Desflurane Group, n=20]: Anaesthesia will be induced with Propofol administered using the automated CLADS and will be maintained with Desflurane.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to the type of anaesthesia intervention.The attending anaesthesiologist will however not be blinded to the technique utilized to administer GA and recovery immediately after extubation inside the OR. The postoperative patient recovery profile will be evaluated by an independent assessor blinded to the technique of GA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLADS group (Active Comparator): Anesthesia will be induced with Propofol administered by CLADSwhich will be set to deliver Propofol according to lean body weight (LBW). A BIS-value of 50 will be used as the target for induction of anesthesia. Thereafter anaesthesia maintenance will be done with Propofol, with the dosing based on adjusted body weight (ABW), and administration controlled with CLADS tuned to consistent anaesthetic depth (BIS-50) feedback from the patients.
  Interventions: Drug: Propofol
- Desflurane group (Active Comparator): Anesthesia will be induced with Propofol administered by CLADSwhich will be set to deliver Propofol according to lean body weight (LBW). A BIS-value of 50 will be used as the target for induction of anesthesia.Thereafter anaesthesia maintenance will be done with desflurane using an agent specific vaporiser, whose dial concentration will be adjusted to maintain a BIS of 50-55 in all the patients
  Interventions: Drug: Propofol; Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — Propofol delivery will be controlled using automated closed loop anaesthesia delivery system which will control propofol delivery rate to consistent anaesthetic depth (BIS-50) feedback from the patient.
Drug: Desflurane — Desflurane delivery will be controlled using a agent specific vaporiser. The dial concentration of the vaporiser will be adjusted to maintain a BIS of 50-55 in the patients.
  Arms: Desflurane group

SUMMARY:
Complete recovery from anaesthesia is absolutely desirable in the obese patients to avoid postoperative airway, oxygen ventilation or sleep apnea related complications. Over the years, Desflurane has emerged as the anaesthetic agent of choice for maintenance of anaesthesia in obese patients for its efficient elimination profile and ability to facilitate early recovery from anaesthesia. Alternatively, Propofol is a commonly used intravenous anesthetic agent administered as a part of total intravenous anesthesia (TIVA) regimen. However, it is a lipid soluble drug and there are concerns that it may accumulate in obese patients due to their increased proportion of body fat Therefore, Propofol TIVA is likely to result in a prolonged duration of action and consequently, delayed emergence from anaesthesia and a protracted recovery time. A recent advance in the delivery of Propofol to the patient is the development of computer-controlled anesthesia delivery systems. These devices deliver Propofol based on feedback from patient's frontal cortex electrical activity as determined by monitoring bispectral index (BIS). Evaluation of anesthesia delivery by these systems has shown that Propofol and maintain depth of anesthesia with far more precision as compared to manual/simple infusion administration. This, in turn, holds promise that recovery from Propofol anaesthesia can also be favourable in the obese patients. An indigenously developed computer-controlled anesthesia delivery sytem is the closed loop anaesthesia delivery system (CLADS), which has been extensively evaluated in patients belonging to different surgical settings. The evidence generated with Propofol anaesthesia delivered by CLADS has shown significant improvement in recovery outcome.The performance of CLADS has not yet been evaluated in obese surgical patients. We hypothesise that in the obese patients undergoing bariatric surgery, automated delivery of Propofol using CLADS would allow precision control of anaesthesia depth, intra-operative haemodynamics, and rapid recovery from anaesthesia. We plan to conduct a randomised controlled investigation to compare patient recovery profile following Desflurane anaesthesia versus CLADS empowered Propofol anaesthesia.

DETAILED DESCRIPTION:
After Institutional Ethics Committee approval and written informed consent, forty-participants (20 per group) aged 18-65 years, ASA physical status I/III, BMI >35-kg/m2, of either sex, and undergoing laparoscopic/robotic bariatric surgery (sleeve gastrectomy or gastric bypass) will be included in this single center (Sir Ganga Ram Hospital, New Delhi-110060, India) prospective, double-blinded, two-arm, randomised controlled study.

The patients who qualify inclusion criteria and consent for recruitment will be randomly divided into one of the two groups:

Group-1 [CLADS Group, n=20]: Anaesthesia will be induced and maintained with Propofol administered using the automated CLADS.

Group-2 [Desflurane Group, n=20]: Anaesthesia will be induced with Propofol administered using the automated CLADS and will be maintained with Desflurane.

Sample-size Estimation

In a previous study, the time-to-eye opening with Desflurane and Propofol was 4.2 minutes and 10.7 minutes, respectively. Based on above, a samples size of 15-patients will be required per group to provide 90% power with a bilateral α-risk value of 0.05 to posit a significant difference in time-to-eye opening. We plan to recruit a total of 40-patients to cover up for unanticipated losses after the recruitment.

Randomization, Allocation Concealment

The patients will be randomly allocated to one of the two groups based on a computer-generated random number table (url:stattrek.com/statistics/random-number-generator.aspx). Randomization sequence concealment will include opaque-sealed envelopes with alphabetic codes whose distribution will be in control of an independent analyst. The envelopes will be opened; patient's data-slip will be pasted on them, and will be sent back to the control analyst.

Blinding Strategy

The attending anaesthesiologist will not be blinded to the technique utilized to administer GA and recovery immediately after extubation inside the OR. However, the postoperative patient recovery profile will be evaluated by an independent assessor blinded to the technique of GA.

Management of Anesthesia

Two peripheral venous lines (18G/20G catheter) will be secured. Standard monitoring (EKG, NIBP, pulse oximeter, EtCO2) will be applied. A BIS sensor (Covidien IIc, Mansfield, USA) will be applied over the patient's forehead according to manufacturer's instruction prior to induction of anaesthesia for monitoring depth of anaesthesia. The BIS monitoring module (Model DSC-XP, Aspect medical system, USA) will facilitate monitoring of anaesthesia depth.

Anaesthesia Technique

All the patients will be administered pre-induction fentanyl-citrate analgesia as per a predefined strategy (total 2-µg/kg IV: 1-µg/kg at 0 minute and 3-minute time point). Pre-oxygenation will be initiated at 3-minute time point or prior to that if there is a fall in oxygen saturation (< 94 percent). In both the groups, at 6-minute time point, anesthesia will be induced with Propofol administered by CLADS. In both the groups CLADS will be set to deliver Propofol according to lean body weight (LBW). A BIS-value of 50 will be used as the target for induction of anesthesia. After induction of anesthesia, atracurium besylate 0.05-mg/kg will be administered for skeletal muscle relaxation to facilitate tracheal intubation. Ventilator settings of CMV, tracheal tube size [7.5-mm I.D (male), 6.5-mm I.D (female)], and breathing circuit (circle-CO2 absorber system) will be the standardized in all the patients. Thereafter, the patients in the CLADS group will receive anaesthesia maintenance with Propofol, with the dosing based on adjusted body weight (ABW), and administration controlled with CLADS tuned to consistent anaesthetic depth (BIS-50) feedback from the patients. The patients in Desflurane group will receive anaesthesia maintenance with Desflurane dial concentration titrated to maintain a BIS of 50-55 in all the patients. Oxygen-air mixture (FiO2 0.50) will be used for ventilation in both the groups.

In addition, starting post-intubation, all the patients will receive 1.0-µg/kg/hr fentanyl infusion for intraoperative analgesia. Intraoperative muscle relaxation will be maintained using atracurium boluses controlled by train-of-four response on peripheral neuromuscular monitor (Infinity TridentNMT Smartpod, Draeger Medical Systems, Inc Telford, USA).

Thirty minutes before the end of surgery, non-opioid analgesics, such as paracetamol 1-gm, and tramadol 100-mg will be administered to the patient. The Propofol or Desflurane delivery will be stopped at the point of completion of skin closure. Residual neuromuscular blockade (assessed with train-of-four response) will be reversed with neostigmine (50-µg/kg) and glycopyrrolate (20-µg/kg).

Thirty minutes before the end of surgery, non-opioid analgesics, such as paracetamol 1-gm, and tramadol 100-mg will be administered to the patient. The Propofol or Desflurane delivery will be stopped at the point of completion of skin closure. Residual neuromuscular blockade (assessed with train-of-four response) will be reversed with neostigmine (50-µg/kg) and glycopyrrolate (20-µg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18-65 years
* BMI > 35 kg/m2
* Either sex
* ASA physical status II & III
* Undergoing laparoscopic/ robotic bariatric surgery

Exclusion Criteria:

* Uncompensated cardiovascular disease (e.g. uncontrolled hypertension, atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance, diastolic dysfunction)
* Hepato-renal insufficiency
* Uncontrolled endocrinology disease (e.g. diabetes mellitus, hypothyroidism)
* Known allergy/hypersensitivity to the study drug
* Pulmonary dysfunction (obstructive/restrictive lung disease)
* Acute/chronic drug dependence/substance abuse
* Requirement of postoperative ventilation
* Refusal to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Early Recovery | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early Recovery | From end of anaesthesia till 30-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Early recovery | From end of anaesthesia till 30-minutes postoperatively
  Ability of the patient to comprehend instructions for shifting himself/herself from the OR table to the transport bed will be assessed using a 4-point scale
Intermediate recovery | From end of anaesthesia till 180-minutes postoperatively
  Time taken to achieve a modified Aldrete score of 9 or 10

SECONDARY OUTCOMES:
Changes in intra-operative heart rate (beats per minute) | From beginning of anesthesia (0-hours, baseline) till 6 hours intra-operatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative blood pressure - systolic , diastolic, and mean (mmHg) | From beginning of anesthesia (0-hours, baseline) till 6 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Postoperative Sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale (OASS)
Postoperative Nausea and Vomiting | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using PONV Scale
Postoperative Analgeisa | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using 10-point Visual Analogue Scale (VAS) Score
Patient Satisfaction | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using a 10-point numeric rating scale
Anesthesia Depth Consistency | From beginning of anaesthesia (0-hours, baseline) till 6 hours intraoperatively]
  Determined by the percentage of the total anaesthesia time in which the BIS scores remain within a score of 10% of the target BIS (i.e. BIS-50) and Varvel criteria parameters; median performance error (MDP), median absolute performance error (MDAPE), wobble and global score

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD, PhD, Study Chair — Post Graduate Institute of Medical Education & Research, Chandigarh, India; Jayashree Sood, MD,FFRCA, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided